CLINICAL TRIAL: NCT07252531
Title: European Investigation of the BrioVAD Left Ventricular Assist System for the Treatment of Refractory Left Ventricular Heart Failure
Brief Title: European Study of the BrioVAD Heart Pump for Advanced Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BrioHealth BV (Industry)
Collaborators: Meditrial SrL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC-04930
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Refractory Heart Failure; Cardiovascular Diseases (CVD)
Keywords: BrioVAD System; Left Ventricular Assist Device
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Device: LVAD implantation

INTERVENTIONS:
Device: LVAD implantation — Implantation of an LVAD in the chest

SUMMARY:
This clinical investigation evaluates the safety and clinical performance of the BrioVAD Left Ventricular Assist System in patients with advanced, refractory left ventricular heart failure who require mechanical circulatory support.

DETAILED DESCRIPTION:
This clinical investigation is conducted to assess the clinical performance and safety of the BrioVAD Left Ventricular Assist System (BrioVAD System) when used for mechanical circulatory support in patients with advanced, refractory left ventricular heart failure.

The BrioVAD System is a fully magnetically levitated, centrifugal-flow left ventricular assist device (LVAD) intended to provide short-term and long-term mechanical circulatory support (MCS) in patients with advanced, refractory heart failure who remain symptomatic despite optimal medical and device therapy. The BrioVAD System is intended for use both inside and outside the hospital environment.

This investigation is designed as a prospective, multi-centre, single-arm, non-inferiority clinical investigation. The performance of the BrioVAD System will be evaluated against a pre-defined Objective Performance Goal (OPG) based on contemporary LVAD clinical outcomes.

The primary objective is to demonstrate that the BrioVAD System provides non-inferior clinical benefit, as measured by survival free from device replacement/removal due to device malfunction at 6 months post-implant, compared with the OPG.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient is ≥ 18 years of age.
2. Patient has a body surface area (BSA) ≥ 1.2 m2.
3. Patient is classified as NYHA Class IV with advanced heart failure refractory to advanced heart failure management or NYHA Class III with dyspnea upon mild physical activity.
4. Patient has a left ventricular ejection fraction (LVEF) ≤ 25% or LVEF < 30% on inotropes or temporary mechanical circulatory support (MCS).
5. Patient is inotrope dependent, OR has a cardiac index (CI) ≤ 2.2 liters/min/m2, while not on inotropes, and also meets one of the following criteria:

   1. Is on optimal medical management (OMM), based on current heart failure practice guidelines for at least 45 out of the last 60 days and is failing to respond or is not able to tolerate OMM; or
   2. Has advanced heart failure for at least 14 days and is dependent on an intra-aortic balloon pump (IABP) or temporary mechanical circulatory support device (MCSD) for at least seven days.
6. Patient has provided voluntary and informed consent.
7. Females of childbearing age agree to use adequate contraception and have a negative pregnancy test.

EXCLUSION CRITERIA:

1. Patient's heart failure etiology is related to restrictive or constrictive physiology (e.g., nondilated hypertrophic cardiomyopathy, cardiac amyloidosis/senile or other infiltrative disease), complex congenital heart disease (e.g., transposition of the great vessels), uncorrected thyroid disease, and/or pericardial disease.
2. Patient had a myocardial infarction within seven days of study enrollment.
3. Patient had cardiothoracic surgery within 30 days of implant with the exception of a procedure to implant temporary MCS: Impella 5.5, Impella CP, or TandemHeart.
4. Patient has physiological conditions or comorbidities which pose high surgical risk or obstacles as determined by the Investigator.
5. Patient has contraindications to warfarin anticoagulation.
6. Patient has known hypo- or hypercoagulable state [e.g., disseminated intravascular coagulation (DIC)], or has a positive heparin-induced thrombocytopenia (HIT) assay and positive serotonin release assay or requires use of a non-heparin alternative anticoagulation strategy for cardiopulmonary bypass in the judgement of the Investigator.
7. Patient is on durable MCS (e.g., LVAD or RVAD).
8. Planned need for durable or temporary RVAD support concomitant with LVAD implant.
9. Patient is on any form of pre-implant temporary MCS other than isolated LVAD support with an intra-aortic balloon pump, Impella 5.5, Impella CP, or TandemHeart.
10. Patient is on any form of pre-implant temporary MCS with a serum lactate dehydrogenase greater than 2.5 times the upper limits of normal or with plasma free hemoglobin > 40 g/dL.
11. Patient has a history of organ transplantation.
12. Patient has a mechanical aortic valve that may not be converted to a bioprosthetic valve at the time of VAD implant.
13. Patient has a platelet count < 50 k/µl.
14. Patient has a history of confirmed untreated abdominal aortic aneurysm (AAA) > 5 cm in diameter.
15. Patient has moderate or severe aortic insufficiency that will not be corrected during the VAD implant procedure.
16. Patient has an uncontrolled systemic infection.
17. Patient has a positive COVID 19 test within 21 days of study enrollment and at least one high risk feature including need for supplemental oxygen or ferritin >1000 ug/L.
18. Patient has severe end-organ dysfunction as evidenced by one or more of the following criteria:

    1. Total bilirubin > 3.0 mg/dL or cirrhosis confirmed by liver imaging or hemodynamic assessment with or without biopsy confirmation.
    2. International normalized ratio (INR) ≥ 2.0 or PTT > 2.5 times control that is not related to anticoagulation therapy.
    3. Glomerular filtration rate (GFR) < 30 mL/ min/1.73 m2 or need for renal replacement therapy.
    4. Severe pulmonary arterial hypertension with a pulmonary vascular resistance (PVR) ≥ 8 Wood units that is not acutely reversible with pharmacologic intervention.
    5. Severe chronic obstructive pulmonary disease (COPD) or restrictive lung disease requiring home oxygen or an FEV1/FVC < 0.7 and FEV1 < 40% predicted.
    6. Mechanical ventilation for more than three days present at the time of study enrollment.
    7. Documented history of pulmonary embolism or pulmonary infarct within 60 days of study enrollment.
    8. History of stroke within 90 days of study enrollment or history of stroke with a mRS ≥ 3 at the time of study enrollment.
    9. Symptomatic cerebrovascular disease and/or uncorrected carotid stenosis > 80%.
    10. Significant peripheral vascular disease (PVD) accompanied by pain at rest or extremity ulceration.
    11. Pre-albumin < 15 mg/dL and/or albumin < 2.5 g/dL.
19. Patient has a non-cardiac comorbidity or illness that would limit survival to less than two years.
20. Patient has a psychiatric disease or disorder, or irreversible cognitive dysfunction, and/or insufficient social support or a history of non-adherence with medical instructions that is likely to impair study compliance.
21. Patient is participating in an interventional clinical trial that may impact or confound the results of the BrioVAD Trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate at 6 months | From enrollment to 6 months on device support

IPD SHARING:
Plan to Share IPD: Undecided